CLINICAL TRIAL: NCT01203969
Title: Safety and Efficacy of Single Port Laparoscopic Surgery in Colon Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kyunghee University Medical Center (Other)
Responsible Party: Principal Investigator, Byung Mo Kang, Clinical Assistant Professor, Kyunghee University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KHNMC IRB 2010-007
Record Dates: First submitted 2010-09-15; First posted 2010-09-17 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-02

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms

ARMS (2):
- Single port laparoscopic surgery (Experimental)
  Interventions: Procedure: Single port laparoscopic surgery
- Conventional laparoscopic surgery (Active Comparator)
  Interventions: Procedure: Conventional laparoscopic surgery

INTERVENTIONS:
Procedure: Single port laparoscopic surgery — laparoscopic surgery in which all the instrument was entered into the abdominal cavity through the single port in the umbilicus
  Arms: Single port laparoscopic surgery
Procedure: Conventional laparoscopic surgery — laparoscopic surgery in which each of the instrument were entered into the abdominal cavity through the multiple port in multiple quadrants of abdomen
  Arms: Conventional laparoscopic surgery

SUMMARY:
This randomized trial is designed to identify the safety and efficacy of single port laparoscopic surgery in colon cancer compared with conventional laparoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

* pathologic proven colon cancer

Exclusion Criteria:

* Tumor located in distal transverse colon, splenic flexure, and descending colon
* distant metastasis
* acute obstruction and/or perforation
* associated with FAP or HNPCC
* synchronous malignancy
* ASA score 3 or 4
* pregnancy
* no consent

Max Age: 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2010-06; Primary Completion 2011-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
rate of intraoperative complication | 1 day
rate of 30 day morbidity and mortality | 1 month

SECONDARY OUTCOMES:
operation time | 1 day
  operative time
degree of postoperative pain | 5 days
  postoperative pain score using visual analog scale (VAS)
amount of postoperative analgesics usage | 5 days
postoperative functional recovery | 7 days
  time to first passage of flatus time to start diet
Duration of postoperative hospital stay | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Suk Hwan Lee, MD. PhD, Principal Investigator — Kyung Hee University School of Medicine
Locations (1):
- Kyung Hee University School of Medicine, Neo Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Kang BM, Park SJ, Lee KY, Lee SH. Single-Port Laparoscopic Surgery Can Be Performed Safely and Appropriately for Colon Cancer: Short-Term Results of a Pilot Randomized Controlled Trial. J Laparoendosc Adv Surg Tech A. 2017 May;27(5):501-509. doi: 10.1089/lap.2016.0467. Epub 2017 Jan 6. PMID 28061037